CLINICAL TRIAL: NCT00982488
Title: Dasatinib in Chronic Myelogenous Leukemia or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemic Subjects Who Are Experiencing Clinical Benefit on Current START or CA180-039 Protocols: Long Term Safety and Efficacy Analysis
Brief Title: Long-term Safety of Dasatinib in Patients With Chronic Myelogenous Leukemia or Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Acronym: START rollover
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-188; 2007-003624-37
Record Dates: First submitted 2009-09-16; First posted 2009-09-23 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Dasatinib; src-Family Kinases; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dasatinib, 50 mg QD to 120 mg BID, Chronic phase (Other): Participants with chronic phase disease continued on the previous study dose of dasatinib, ranging from 50 mg once daily (QD) to 120 mg twice daily (BID).
  Interventions: Drug: Dasatinib
- Imatinib, 400 mg BID, Chronic phase (Other): Participants with chronic phase disease received 400 mg of imatinib twice BID.
  Interventions: Drug: Imatinib
- Dasatinib, 50 mg QD to 120 mg BID, Advanced phase, AP (Other): Participants with advanced phase disease, accelerated phase (AP), continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID.
  Interventions: Drug: Dasatinib
- Dasatinib, 50 mg QD to 120 mg BID, Advanced phase, MBP (Other): Participants with advanced phase disease, myeloid blast cell (MBP), continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID.
  Interventions: Drug: Dasatinib
- Dasatinib, 50 mg QD to 120 mg BID, Advanced phase, Ph+ ALL (Other): Participants with advanced phase disease, Philadelphia chromosome positive acute lymphoblastic leukemia (Ph+ ALL), continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Dasatinib was supplied as 20- and 50-mg tablets.
  Other Names: BMS-354825; Sprycel; Src Kinase
  Arms: Dasatinib, 50 mg QD to 120 mg BID, Advanced phase, AP; Dasatinib, 50 mg QD to 120 mg BID, Advanced phase, MBP; Dasatinib, 50 mg QD to 120 mg BID, Advanced phase, Ph+ ALL; Dasatinib, 50 mg QD to 120 mg BID, Chronic phase
Drug: Imatinib — Imatinib was supplied as 100- and 400-mg tablets.
  Other Names: Gleevec/Glivec
  Arms: Imatinib, 400 mg BID, Chronic phase

SUMMARY:
This study assesses the long-term safety and tolerability of dasatinib administered to patients with chronic myelogenous leukemia or Philadelphia chromosome positive acute lymphoblastic leukemia and experienced clinical benefit from treatment with dasatinib or imatinib in previous protocols.

ELIGIBILITY:
Key Inclusion Criteria

* Signed written informed consent
* Received treatment in protocols CA180-005, CA180-006, CA180-013, CA180-015 or CA180-017, or CA180-039
* Received clinical benefit with dasatinib or imatinib (study CA180017) in the opinion of the Investigator
* Men and women, ages 18 and older

Key Exclusion Criteria

* A serious uncontrolled medical disorder or active infection that would impair the ability of the patient to receive protocol therapy
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
* Patients currently taking drugs, including but not limited to quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycins, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, ziprasidone, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, and lidoflazine, which are generally accepted to have a risk of causing Torsades de Pointes
* Patients taking medications known to be potent CYP3A4 inhibitors (ketoconazole, ritonavir) or inducers (rifampin, efavirenz)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2007-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (69):
- United States (17):
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Ucla Department Of Medicine, Los Angeles, California
  - Stanford University School Of Medicine, Stanford, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University Of Chicago, Chicago, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - University Of Kansas Medical Center, Westwood, Kansas
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - University Of Michigan Medical Center, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Oregon Health & Sci Univ, Portland, Oregon
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Ut Southwestern Medical Center At Dallas, Dallas, Texas
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
- Local Institution, Adelaide, South Australia, Australia
- Local Institution, Mont-godinne, Belgium
- Brazil (4):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Campinas, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (2):
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- Local Institution, Helsinki, Finland
- France (7):
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (3):
  - Local Institution, Hamburg
  - Local Institution, Leipzig
  - Local Institution, Mannheim
- Local Institution, Budapest, Hungary
- Local Institution, Dublin, Dublin, Ireland
- Local Institution, Ramat Gan, Israel
- Italy (4):
  - Local Institution, Bologna
  - Local Institution, Napoli
  - Local Institution, Orbassano (to)
  - Local Institution, Roma
- Local Institution, Trondheim, Norway
- Local Institution, Lima, Lima Province, Peru
- Poland (5):
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Warsaw
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- South Africa (2):
  - Local Institution, Groenkloof, Gauteng
  - Local Institution, Parktown, Gauteng
- South Korea (2):
  - Local Institution, Jeollanam-do
  - Local Institution, Seoul
- Local Institution, Barcelona, Spain
- Sweden (5):
  - Local Institution, Gothenburg
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Umeå
  - Local Institution, Uppsala
- Local Institution, Basel, Switzerland
- Local Institution, Bangkok, Thailand
- United Kingdom (3):
  - Local Institution, London, Greater London
  - Local Institution, Glasgow, Scotland
  - Local Institution, Newcastle, Tyne and Wear

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 238 patients were enrolled: 200 with chronic phase chronic myelogenous leukemia (CML) and 38 with advanced phase disease (34 with acclelerated phase CML, 3 with myeloid blast phase CML, and 1 with Philadelphia chromosome positive acute lymphoblastic leukemia.) All but 1 CML patient, who no longer met study criteria, received treatment.
Groups:
- Dasatinib 50 mg QD to 120 mg BID, Chronic Phase: Participants with chronic phase disease were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg once daily (QD) to 120 mg twice daily (BID). Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Imatinib, 400 mg BID, Chronic Phase: Participants chronic phase disease received 400 mg of imatinib BID. Dose reduction to 600 mg/day (300 mg BID) was permitted, provided the participant had not previously received that dose prior to entry into CA180-017. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP: Participants with advanced phase disease, accelerated phase (AP) were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID . Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MPB: Participants with advanced phase disease, myeloid blast phase (MPB), were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID . Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, Ph+ ALL: Participants with advanced phase disease, Philadelphia chromosome positive acute lymphoblastic leukemia (Ph+ ALL), were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID . Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
Period: Overall Study
Arm/Group | Dasatinib 50 mg QD to 120 mg BID, Chronic Phase | Imatinib, 400 mg BID, Chronic Phase | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MPB | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, Ph+ ALL
Started | 185 (Received treatment) | 14 (Received treatment) | 34 (Received treatment) | 3 (Received treatment) | 1 (Received treatment)
Completed | 0 (Still receiving treatment) | 0 (Still receiving treatment) | 0 (Still receiving treatment) | 0 (Still receiving treatment) | 0 (Still receiving treatment)
Not Completed | 185 | 14 | 34 | 3 | 1
Not completed — Administrative reason by sponsor | 81 | 3 | 11 | 0 | 0
Not completed — Adverse event unrelated to study drug | 5 | 1 | 0 | 0 | 0
Not completed — Death | 11 | 0 | 2 | 0 | 0
Not completed — Disease progression | 30 | 5 | 10 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 1 | 1 | 1 | 0 | 0
Not completed — Other | 15 | 1 | 3 | 1 | 0
Not completed — Poor compliance/noncompliance | 0 | 1 | 0 | 0 | 0
Not completed — Stem cell transplant | 2 | 0 | 0 | 1 | 0
Not completed — Study drug toxicity | 34 | 1 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Imatinib, 400 mg BID, Chronic Phase: Participants with chronic phase disease received 400 mg of imatinib BID. Dose reduction to 600 mg/day (300 mg BID) was permitted, provided the participant had not previously received that dose prior to entry into CA180-017. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP: Participants with advanced phase disease, accelerated phase (AP), were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID . Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Total: Total of all reporting groups
Arm/Group | Dasatinib 50 mg QD to 120 mg BID, Chronic Phase | Imatinib, 400 mg BID, Chronic Phase | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MPB | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, Ph+ ALL | Total
Number analyzed (Participants) | 185 | 14 | 34 | 3 | 1 | 237
Age, Customized [Number; unit: Participants]
  Younger than 21 years | 0 | 0 | 0 | 0 | 0 | 0
  21-45 years | 46 | 5 | 7 | 0 | 0 | 58
  46-65 years | 88 | 5 | 17 | 3 | 1 | 114
  66-75 years | 40 | 3 | 9 | 0 | 0 | 52
  Older than 75 years | 11 | 1 | 1 | 0 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 6 | 15 | 2 | 1 | 115
  Male | 94 | 8 | 19 | 1 | 0 | 122
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 167 | 10 | 26 | 2 | 1 | 206
  Black/African American | 8 | 0 | 2 | 0 | 0 | 10
  Asian | 7 | 1 | 6 | 0 | 0 | 14
  Other | 3 | 3 | 0 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died and Had Serious Adverse Events (SAEs), Related SAEs, Adverse Events (AEs) Leading to Discontinuation, Related AEs Leading to Discontinuation, Related AEs, and Related AEs of Special Interest
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=drug-related; having certain, probable, possible, or unknown relationship to study drug.
Time Frame: Day 1 of treatment through a maximum of 82 months + 30 days
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Groups:
- Dasatinib, 50 mg QD to 120 mg BID, Chronic Phase: Participants with chronic phase disease were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg once daily (QD) to 120 mg twice daily (BID). Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Imatinib, 400 mg BID, Chronic Phase: Participants with chronic phase disease received 400 mg of imatinib twice daily (BID). Dose reduction to 600 mg/day (300 mg BID) was permitted, provided the participant had not previously received that dose prior to entry into CA180-017. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MBP: Participants with advanced phase disease, myeloid blast phase (MBP), were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID . Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
Arm/Group | Dasatinib, 50 mg QD to 120 mg BID, Chronic Phase | Imatinib, 400 mg BID, Chronic Phase | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MBP | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, Ph+ ALL
Number analyzed (Participants) | 185 | 14 | 34 | 3 | 1
Participants
  All deaths | 22 | 0 | 4 | 0 | 0
  Deaths within 30 days of last dose | 9 | 0 | 2 | 0 | 0
  SAEs | 57 | 3 | 15 | 1 | 1
  Drug-related SAEs | 28 | 2 | 9 | 0 | 0
  AEs leading to discontinuation | 39 | 1 | 10 | 0 | 1
  Drug-related AEs leading to discontinuation | 29 | 1 | 8 | 0 | 0
  Drug-related AEs | 140 | 7 | 27 | 2 | 0
  Drug-related AEs of special interest | 111 | 4 | 20 | 1 | 0

ADVERSE EVENTS:
Groups:
- Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP: Participants with advanced phase disease, accelerated phase (AP), were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID. Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MBP: Participants with advanced phase disease, myeloid blast phase (MBP), were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID. Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
- Dasatinib, 50 mg QD to 120 mg, Advanced Phase, Ph+ ALL: Participants with advanced phase disease, Philadelphia chromosome positive acute lymphoblastic leukemia (Ph+ ALL), were rolled over from previous studies CA180-039, CA180-043, and the SRC/ABL tyrosine kinase inhibition activity: Research trials (START). Participants continued on the previous study dose of dasatinib, ranging from 50 mg QD to 120 mg BID. Dose escalations to optimize response and dose reductions for toxicity were permitted. Participants received study medication until disease progression, unacceptable toxicity, failure to serve patient's best interest, withdrawal of consent, or study closure.
Arm/Group | Dasatinib, 50 mg QD to 120 mg BID, Chronic Phase | Imatinib, 400 mg BID, Chronic Phase | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MBP | Dasatinib, 50 mg QD to 120 mg, Advanced Phase, Ph+ ALL
Serious Adverse Events (participants affected / at risk) | 57/185 | 3/14 | 15/34 | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 138/185 | 10/14 | 24/34 | 2/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 50 mg QD to 120 mg BID, Chronic Phase (N=185) | Imatinib, 400 mg BID, Chronic Phase (N=14) | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP (N=34) | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MBP (N=3) | Dasatinib, 50 mg QD to 120 mg, Advanced Phase, Ph+ ALL (N=1)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Oophorectomy bilateral (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Effusion (General disorders) | 1 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 1 | 3 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 0 | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Elderly (Social circumstances) | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 0 | 3 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 2 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 50 mg QD to 120 mg BID, Chronic Phase (N=185) | Imatinib, 400 mg BID, Chronic Phase (N=14) | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, AP (N=34) | Dasatinib, 50 mg QD to 120 mg BID, Advanced Phase, MBP (N=3) | Dasatinib, 50 mg QD to 120 mg, Advanced Phase, Ph+ ALL (N=1)
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 13 | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 1 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 25 | 1 | 4 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 31 | 0 | 4 | 0 | 0
Viral infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 1 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 9 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 12 | 0 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 67 | 1 | 17 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 19 | 2 | 2 | 1 | 0
Face oedema (General disorders) | 2 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 25 | 1 | 3 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 0 | 1 | 1 | 0
Blood fibrinogen decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 0 | 5 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 1 | 3 | 0 | 0
Pyrexia (General disorders) | 15 | 1 | 1 | 0 | 0
Blood bilirubin (Investigations) | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 0 | 4 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 0 | 2 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 14 | 1 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.